CLINICAL TRIAL: NCT00587834
Title: A Clinical Trial to Evaluate Gintuit (TM) (Allogeneic Cultured Keratinocytes and Fibroblasts in Bovine Collagen) as an Alternative to Tissue From the Palate to Enhance Oral Soft Tissue Regeneration and Wound Healing
Brief Title: Safety and Efficacy of Gintuit(TM)for Oral Soft Tissue Regeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-PER-002-CTX
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Within-subject design: one side of the mouth receives Gintuit
  Interventions: Device: Gintuit
- 2 (Active Comparator): Within-subject control: one side of mouth receives tissue harvested from the palate
  Interventions: Other: Autologous palatal tissue

INTERVENTIONS:
Device: Gintuit — Application of Gintuit at Day 0 to the gingival bed
  Arms: 1
Other: Autologous palatal tissue — Tissue will be harvested from the subject's palate and placed on the gingival bed
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate Gintuit as a safe and effective alternative to palatal tissue in the treatment of subjects (with recession-type defects) who have an insufficient zone of attached gingiva associated with at least two nonadjacent teeth.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age but no more than 70 years of age.
* Subject has at least two non-adjacent teeth in contralateral quadrants of the same jaw with an insufficient zone (< or = 1mm) of attached gingiva that requires soft tissue grafting. (1-3 teeth may be treated. In case of adjacent teeth requiring grafting, only one tooth at each site will act as test or control tooth, but all teeth will get the same treatment).
* Root coverage is not desired at the time of grafting.
* Females of childbearing potential must have a documented negative urine pregnancy test.
* Subjects must have read, understood and signed an institutional review board (IRB) approved Informed Consent Form.
* Subjects must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

* Subject with class III recession in the presence of a shallow vestibule or class IV recession.
* Subject with vestibule depth of less than 7mm from base of recession.
* Subject with any systemic conditions that could compromise wound healing and preclude periodontal surgery (i.e., diabetes mellitus, cancer, human immunodeficiency virus (HIV), bone metabolic diseases).
* Subject who is currently receiving or has received within two months prior to study entry, systemic corticosteroids, immunosuppressive agents, radiation therapy, and/or chemotherapy which could compromise wound healing and preclude periodontal surgery.
* Subject with the presence of acute infectious lesions in the areas intended for surgery.
* Subject who has used any tobacco product within 3 months.
* Subject who is taking intramuscular or intravenous bisphosphonates.
* Subject with only molar teeth suitable for soft tissue grafting.
* Subject with teeth that have Miller Grade 2 or higher mobility.
* Subject with known hypersensitivity to bovine collagen and/or iodine (shellfish allergy).
* Subject who has received an investigational drug or biological/bioactive treatment within 30 days prior to study enrollment (medical or dental).
* Subject who was previously treated with Gintuit, Dermagraft or any other skin graft at the target site(s) or immediately adjacent teeth.
* Subject, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGuire, DDS, Principal Investigator — Perio Health Professionals, PLLC
Locations (4):
- United States (4):
  - Nevins Perio, LLC, Boston, Massachusetts
  - Michigan Center for Oral Health Research, Ann Arbor, Michigan
  - Perio Health Professionals, PLLC, Houston, Texas
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas

REFERENCES:
- [Result] McGuire MK, Scheyer ET, Nevins ML, Neiva R, Cochran DL, Mellonig JT, Giannobile WV, Bates D. Living cellular construct for increasing the width of keratinized gingiva: results from a randomized, within-patient, controlled trial. J Periodontol. 2011 Oct;82(10):1414-23. doi: 10.1902/jop.2011.100671. Epub 2011 Mar 29. PMID 21513473

RESULTS

PARTICIPANT FLOW:
Groups:
- Gintuit and Autologous Free Gingival Graft (FGG): Single application of Gintuit and FGG (control); split-mouth design
Period: Overall Study
Arm/Group | Gintuit and Autologous Free Gingival Graft (FGG)
Started | 96
Completed | 96
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gintuit and Autologous Free Gingival Graft (FGG)
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 47.14 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 85
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 87
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least 2 mm Keratinized Tissue (KT) at 6 Months at the Gintuit Treated Site.
Description: The superiority of Gintuit relative to a pre-defined standard (50% success) for a 2 mm KT threshold after six months.
Time Frame: 6 months
Population: Per protocol the first 2 subjects per Investigator were training subjects and evaluated for safety only. There were 11 training subjects and the remaining 85 subjects were analyzed for all efficacy outcomes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Gintuit: Single application;split-mouth design
Arm/Group | Gintuit
Number analyzed (Participants) | 85
percentage of participants | 95.3 [88.4 to 98.7]
Statistical Analysis 1: Comparison: Gintuit; Superiority relative to a pre-defined standard (50% success); Test type: Superiority or Other; p < 0.0001, Exact Bionomial Test

2. Secondary Outcome: Color Same as Adjacent Tissues After 6 Months (Superiority)
Description: An examiner assessed color of both treated sites compared with the adjacent, non-treated tissue. The assessment was recorded as "More Red", "Equally Red", or "Less Red" as compared to adjacent, non-treated tissue. A match in color with the surrounding tissue is considered a positive aesthetic outcome.
Time Frame: 6 months
Population: See description in primary outcome measure.
Measure: Number; unit: Participants
Groups:
- Gintuit Not Equally Red as Adjacent Tissue: Not Equally Red includes responses of "more red" and "less red"
Arm/Group | Gintuit Equally Red as Adjacent Tissue | Gintuit Not Equally Red as Adjacent Tissue
Number analyzed (Participants) | 85 | 85
Participants
  Control Equally Red as Adjacent Tissue | 23 | 0
  Control Not Equally Red as Adjacent Tissue | 56 | 6
Statistical Analysis 1: Comparison: Gintuit Equally Red as Adjacent Tissue vs Gintuit Not Equally Red as Adjacent Tissue; Compare participants with (1) Gintuit equally red and Control not equally red to (2) Gintuit not equally red and Control equally red; Test type: Superiority or Other; p < 0.0001, McNemar

3. Secondary Outcome: Texture Same as Adjacent Tissues After 6 Months (Superiority)
Description: An examiner assessed texture of both treated sites compared with the adjacent, non-treated tissue. The assessment was recorded as "More Firm", "Equally Firm", or "Less Firm" as compared to adjacent, non-treated tissue. A match in texture with the surrounding tissue is considered a positive aesthetic outcome.
Time Frame: 6 months
Population: See description in primary outcome measures.
Measure: Number; unit: Participants
Groups:
- Gintuit Not Equally Firm as Adjacent Tissue: Not Equally Firm includes responses of "less firm" and "more firm"
Arm/Group | Gintuit Equally Firm as Adjacent Tissue | Gintuit Not Equally Firm as Adjacent Tissue
Number analyzed (Participants) | 85 | 85
Participants
  Control Equally Firm as Adjacent Tissue | 46 | 0
  Control Not Equally Firm as Adjacent Tissue | 35 | 4
Statistical Analysis 1: Comparison: Gintuit Equally Firm as Adjacent Tissue vs Gintuit Not Equally Firm as Adjacent Tissue; Compare participants with (1)Gintuit equally firm and Control not equally firm to (2) Gintuit not equally firm and Control equally firm; Test type: Superiority or Other; p < 0.0001, McNemar

4. Secondary Outcome: Percentage of Subjects With at Least 1 mm Keratinized Tissue (KT) at 6 Months at the Gintuit Treated Site.
Description: The superiority of Gintuit relative to a pre-defined standard (80% success) for a 1 mm KT threshold after six months.
Time Frame: 6 months
Population: See description in primary outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Gintuit
Number analyzed (Participants) | 85
Percentage of Participants | 100 [95.8 to 100.0]
Statistical Analysis 1: Comparison: Gintuit; Superiority relative to a pre-defined threshold (80%) success; Test type: Superiority or Other; p < 0.0001, Exact binomial test

5. Secondary Outcome: Patient Preference After 6 Months/Early Termination (Superiority)
Description: Number of patients expressing preference for Gintuit.
Time Frame: 6 months
Population: See description in primary outcome measure.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Gintuit: Single application of Gintuit and FGG (control); split-mouth design. Number of subjects preferring Gintuit over Control.
Arm/Group | Gintuit
Number analyzed (Participants) | 85
participants | 61 [61.0 to 81.0]
Statistical Analysis 1: Comparison: Gintuit; The proportion of Gintuit as the preferred procedure; Test type: Superiority or Other; p < 0.0001, Exact binomial test

6. Secondary Outcome: Surgical Site Sensitivity Mild or Absent After 1 Week(Superiority)
Description: The sensitivity of Gintuit, Free Gingival Graft (FGG) and palatal donation sites was assessed with a puff of air and rated by the Investigator as none, mild, moderate or severe sensitivity. The sensitivity of Control was determined as the most sensitive of FGG and palatal donation sites.
Time Frame: 6 months
Population: See description in primary outcome measures. The presence of Coe-Pak (protective periodontal dressing) at Week 1 prohibited the assessment of sensitivity for 14 subjects. The analysis was performed on 71 of the 85 subjects evaluated for efficacy.
Measure: Number; unit: Participants
Groups:
- Gintuit Not Sensitive: Included ratings of None and Mild
- Gintuit Sensitive: Included ratings of Moderate and Severe
Arm/Group | Gintuit Not Sensitive | Gintuit Sensitive
Number analyzed (Participants) | 71 | 71
Participants
  Control Not Sensitive | 67 | 3
  Control Sensitive | 1 | 0
Statistical Analysis 1: Comparison: Gintuit Not Sensitive vs Gintuit Sensitive; Compare participants with (1) Gintuit not sensitive and Control sensitive to (2) Gintuit sensitive and Control not sensitive; Test type: Superiority or Other; p = 0.3173, McNemar; McNemar's paired comparison test

7. Secondary Outcome: Pain Absent After 3 Days (Superiority)
Description: Pain Assessment(Modified Intent-to-Treat Population)
Time Frame: Day 3
Reporting Status: Not Posted
Measure: Number; unit: Participants

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Gintuit: Adverse events occurring at the Gintuit treated site
- Free Gingival Graft: Adverse events occurring at the autologous free gingival graft site
- Palatal Donation Site: Adverse events occurring at the palatal donation site
- Mouth: Adverse events occurring in the mouth and not localized to the Gintuit, FGG, or palatal donation sites.
- Other: Adverse events occurring at any other location in the body or systemic conditions
Arm/Group | Gintuit | Free Gingival Graft | Palatal Donation Site | Mouth | Other
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96 | 0/96 | 0/96 | 3/96
Other Adverse Events (participants affected / at risk) | 0/96 | 0/96 | 0/96 | 0/96 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gintuit (N=96) | Free Gingival Graft (N=96) | Palatal Donation Site (N=96) | Mouth (N=96) | Other (N=96)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pains (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant Metastatic Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Secondary outcome measures were tested with a closed testing strategy; therefore pain was not tested (no p-value) because previous endpoint (site sensitivity) failed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review communications prior to public release and can embargo communications regarding trial results for at least 30 days in advance of public release. The sponsor can request removal of any confidential or proprietary information provided by sponsor and extend such review period for another 90 days to file patent applications or take other steps to protect the sponsor's intellectual property interests.